CLINICAL TRIAL: NCT00147199
Title: TRIUMPH I: Double Blind Placebo Controlled Clinical Investigation Into the Efficacy and Tolerability of Inhaled Treprostinil Sodium in Patients With Severe Pulmonary Arterial Hypertension
Brief Title: Clinical Investigation Into Inhaled Treprostinil Sodium in Patients With Severe Pulmonary Arterial Hypertension (PAH)
Acronym: TRIUMPH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LRX-TRIUMPH 001
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2013-08-12 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2013-07

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled treprostinil (Experimental): 0.9 mg/mL treprostinil for inhalation supplied in 2.9mL ampoules for use in ultra sonic nebulizer
  Interventions: Drug: Inhaled treprostinil
- Placebo (Placebo Comparator): Placebo inhalation solution for use in ultrasonic nebulizer
  Interventions: Drug: Placebo inhalation solution

INTERVENTIONS:
Drug: Inhaled treprostinil — Doses are titrated to 9 breaths four times daily. Each breath produces an 18 mcg dose of inhaled treprostinil.
  Other Names: Tyvaso
  Arms: Inhaled treprostinil
Drug: Placebo inhalation solution — Doses are titrated to 9 breaths four times daily.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind placebo-controlled clinical investigation into the efficacy and tolerability of inhaled treprostinil in patients with severe pulmonary arterial hypertension. The primary outcome is the change in 6-minute walk distance from baseline to week 12.

DETAILED DESCRIPTION:
Patients who have been on a stable dose of 125 mg twice daily (bid) of bosentan or any stable dose of sildenafil for at least three months prior to study start were randomized to either treprostinil inhalation solution or matching placebo.

Administration of study medication was performed by inhalation with the OPTINEB™ ultrasonic nebulizer.

The proposed dosing regimen was four times daily-upon awakening, at midday, evening (dinner time) and bedtime.

After a patient has completed the twelve-week study period, they were given the option of enrolling into an open-label extension study.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable, pulmonary arterial hypertension diagnosed as either idiopathic or familial PAH, collagen vascular disease associated PAH, HIV PAH, or PAH induced by anorexigens, New York Heart Association (NYHA) Class III or Class IV.
* Been on a stable dose of 125 mg twice daily (bid) of bosentan OR any stable dose of sildenafil for at least three months prior to study start
* An unencouraged six minute walk test (6MWT) of between 200 and 450 meters at screening
* Cardiac catheterization within the past 13 months consistent with PAH, specifically mean pulmonary artery pressure (PAPm) ≥25 mmHg (at rest), pulmonary capillary wedge pressure (PCWP) (or left ventricular end diastolic pressure) ≤15 mmHg, and pulmonary vascular resistance (PVR) >3 mmHg/L/min
* Within the past 12 months, patients must have had a chest radiograph consistent with the diagnosis of PAH
* Willing and able to follow all study procedures

Exclusion Criteria:

* Considering pregnancy, are pregnant and/or lactating
* PAH due to conditions other than noted in the above inclusion criteria.
* Have had any change in or discontinued any PAH medication within the last three months, including but not limited to endothelin receptor antagonist (ERA), or calcium channel blockers (CCB) (with the exception of anticoagulants)
* Have received any prostanoid within the 30 days before screening or are scheduled to receive any during the course of the study
* Have received any investigational medication within 30 days prior to the start of this study or are scheduled to receive another investigational drug during the course of this study
* Have a known intolerance to any drug, especially to treprostinil sodium or prostanoids
* Have an increased risk of hemorrhage
* Have a new type of chronic therapy (e.g., a different category of vasodilator, diuretic) for PAH added within the last month, except anticoagulants
* Have any musculoskeletal disease or any other disease that would limit ambulation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2005-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - UCSD Medical center, La Jolla, California
  - UCLA Medical Center, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Orlando Heart Center, Orlando, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Bethe Israel Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UTSW Medical Center, Dallas, Texas
- Austria (2):
  - Universitatsklinikfur Innere Medizin II, Wein, Vienna
  - Medical University Graz, Graz
- Belgium (2):
  - Universite Libre de Bruxelles, Brussels
  - University Hospital Gasthuisburg, Leuven
- Hospital Antoine Beclere, Paris, France
- Univesitatsklinikum Giessen und Marburg GmbH, Geißen, Germany
- Pulmonary Hypertension Unit, Dublin, Ireland
- Israel (3):
  - Rambam Medical Center, Haifa
  - The Pulmonary Institute, Jerusalem
  - The Pulmonary Institute, Petach Tikvah 49100
- Instituto Malattie dell'Apparato Vascolare, Bologna, Italy
- University of Barcelona, Barcelona, Spain
- United Kingdom (3):
  - Papworth Hospital, Cambridge
  - Scottish Pulmonary Vascular Unit, Glasgow GII 6NT
  - Royal Fee Hospital, London

REFERENCES:
- [Derived] McLaughlin VV, Benza RL, Rubin LJ, Channick RN, Voswinckel R, Tapson VF, Robbins IM, Olschewski H, Rubenfire M, Seeger W. Addition of inhaled treprostinil to oral therapy for pulmonary arterial hypertension: a randomized controlled clinical trial. J Am Coll Cardiol. 2010 May 4;55(18):1915-22. doi: 10.1016/j.jacc.2010.01.027. PMID 20430262
- See also: The mission of the Pulmonary Hypertension Association is to seek a cure, and to provide hope, support and education, and to promote awareness and to advocate for the pulmonary hypertension community. — http://www.phassociation.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 7 June 2005 and the last subject exited the study on 12 Oct 2007.
Groups:
- Inhaled Treprostinil: Initial dose: 3 breaths. Titrated to 9 breaths, four times daily.
- Placebo: Identical placebo inhalation solution
Period: Overall Study
Arm/Group | Inhaled Treprostinil | Placebo
Started | 115 | 120
Completed | 102 | 110
Not Completed | 13 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Treprostinil | Placebo | Total
Number analyzed (Participants) | 115 | 120 | 235
Age, Continuous [Mean (Full Range); unit: years] | 55 (13.1) [20 to 75] | 52 [18 to 75] | 54 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 98 | 191
  Male | 22 | 22 | 44
Pulmonary Arterial Hypertension (PAH) Etiology [Number; unit: participants]
  Idiopathic PAH (IPAH) | 64 | 67 | 131
  Connective Tissue Disease (CTD) | 40 | 37 | 77
  Other | 11 | 16 | 27
Background PAH Therapy [Number; unit: participants]
  Bosentan | 77 | 88 | 165
  Sildenafil | 38 | 32 | 70
Time on Background Therapy [Mean (Standard Deviation); unit: weeks]
  Bosentan | 98 (79) | 90 (75) | 94 (77)
  Sildenafil | 65 (60) | 77 (69) | 70 (64)
Baseline NYHA Class [Number; unit: participants]
  Class III | 112 | 118 | 230
  Class IV | 3 | 2 | 5
Baseline Six-Minute Walk Distance (6MWD) [Mean (Standard Deviation); unit: meters] | 346 (63) | 351 (69) | 348 (66)

OUTCOME MEASURES:

1. Primary Outcome: Peak 6-minute Walk Distance
Description: Change in peak 6-minute walk distance from baseline to Week 12. Peak 6MWD was defined as a 6-minute walk test (6MWT) within 10 to 60 minutes after study drug inhalation
Time Frame: 12 weeks
Population: Intention to treat analysis
Measure: Median (Inter-Quartile Range); unit: meters
Groups:
- Placebo: Initial dose: 3 breaths. Titrated to 9 breaths, four times daily.
Arm/Group | Inhaled Treprostinil | Placebo
Number analyzed (Participants) | 115 | 120
meters
  Week 12 | 366.0 [300.0 to 423.0] | 360.0 [296.0 to 414.9]
  Change from Baseline | 21.6 [-8.0 to 54.0] | 3.0 [-26.0 to 31.5]
Statistical Analysis 1: Comparison: Inhaled Treprostinil vs Placebo; Sample size was calculated based on the primary endpoint; change in 6MWD at Week 12. Assuming a between-treatment difference of 35m, a standard deviation of 75m, and a type I (alpha) error of 0.05 (i.e., two-sided p-value of less than 0.05), in order to have 90% power to detect this difference, 100 subjects per treatment group were required for this trial (total n=200). This allowed for a dropout rate of 10% as 110 subjects per group was planned; Test type: Superiority or Other; p = 0.00044, ANCOVA; Lowest rank was assigned for death, discontinuation due to disease progression, and for patients who initiated additional approved PAH therapy; Hodges-Lehmann Estimate = 20.0, 95% CI 2-sided [8.0 to 32.8]

2. Secondary Outcome: Clinical Worsening Events
Description: Clinical worsening was defined as the first incidence of clinical worsening from randomization to the first occurrence of death, transplantation, hospitalization for PAH, or initiation of additional approved PAH therapy.
Time Frame: 12 weeks
Population: Intention to treat population
Measure: Number; unit: clinical worsening events
Arm/Group | Inhaled Treprostinil | Placebo
Number analyzed (Participants) | 115 | 120
clinical worsening events | 4 | 6

3. Secondary Outcome: Borg Dyspnea Score
Description: The Borg dyspnea score is a patient reported number between 0 (no perceived shortness of breath) and 10 (maximum perceived shortness of breath), obtained at the completion of each 6MWT.
Time Frame: 12 weeks
Population: Intention to treat population. A Week 12 observation was not present for one subject and that data point is not included in the analysis.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Inhaled Treprostinil | Placebo
Number analyzed (Participants) | 115 | 119
score
  Week 12 | 3.68 (2.26) | 3.91 (2.33)
  Change from Baseline | 0.0 (2.07) | 0.0 (1.72)
Statistical Analysis 1: Comparison: Inhaled Treprostinil vs Placebo; Test type: Superiority or Other; p = 0.623, Wilcoxon rank sum test; Hodges-Lehmann (H-L) = 0.0, 95% CI 2-sided [-0.5 to 0.0]

4. Secondary Outcome: New York Heart Association (NYHA) Functional Classification
Description: Change in NYHA functional class at Week 12. NYHA classifications:
  Class I - Patients with pulmonary hypertension but without resulting limitation of physical activity. Ordinary physical activity does not cause undue dyspnea or fatigue, chest pain or near syncope.
  Class II - Patients with pulmonary hypertension resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity causes undue dyspnea or fatigue, chest pain or near syncope.
  Class III - Patients with pulmonary hypertension resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes undue dyspnea or fatigue, chest pain or near syncope.
  Class IV - Patients with pulmonary hypertension in the inability to carry out any physical activity without symptoms. These patients manifest signs of right heart failure. Dyspnea and/or fatigue may even be present at rest. Discomfort is increased by any physical activity.
Time Frame: 12 weeks
Population: Intention to treat population
Measure: Number; unit: participants
Arm/Group | Inhaled Treprostinil | Placebo
Number analyzed (Participants) | 115 | 120
participants
  NYHA Class II | 22 [0 to 0] | 22
  NYHA Class III | 88 | 93
  NYHA Class IV | 5 | 5
Statistical Analysis 1: Comparison: Inhaled Treprostinil vs Placebo; Test type: Superiority or Other; p = 0.807, Wilcoxon rank sum test — Imputation strategies were implemented for 16 inhaled treprostinil subjects and 9 placebo subjects without values reported at Week 12; Hodges-Lehmann (H-L) = 0.0, 95% CI 2-sided [0.0 to 0.0]

5. Secondary Outcome: Trough 6MWD at Week 12
Description: Change in 6MWD from Baseline to trough 6MWD at Week 12. Trough was defined as a 6MWT conducted at least 4 hours following study drug inhalation.
Time Frame: 12 Weeks
Population: Intention to treat population
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Inhaled Treprostinil | Placebo
Number analyzed (Participants) | 115 | 120
meters
  Week 12 trough | 364.0 [313.0 to 420.0] | 365.0 [289.0 to 422.0]
  Change from Baseline | 12.4 [-10.0 to 51.3] | 0.8 [-17.9 to 25.0]
Statistical Analysis 1: Comparison: Inhaled Treprostinil vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA; Hodges-Lehmann (H-L) = 13.7, 95% CI 2-sided [4.0 to 24.8]

6. Secondary Outcome: Peak 6MWD at Week 6
Description: Change in peak 6MWD between Baseline and Week 6.
Time Frame: 6 weeks
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Inhaled Treprostinil | Placebo
Number analyzed (Participants) | 115 | 120
meters
  Week 6 Values | 375 [305 to 421] | 367 [292 to 419]
  Change from Baseline | 21.6 [-4.0 to 51.8] | 3.0 [-16.5 to 22.0]
Statistical Analysis 1: Comparison: Inhaled Treprostinil vs Placebo; Test type: Superiority or Other; p = 0.0003, Wilcoxon rank sum test; Hodges-Lehmann (H-L) = 18.5, 95% CI 2-sided [8.5 to 28.3]

7. Secondary Outcome: Quality of Life (Minnesota Living With Heart Failure)
Description: Quality of life as measured by the Minnesota Living With Heart Failure (MLWHF) questionnaire was evaluated at baseline and at Week 12. The MLWHF questionnaire consists of 21 questions assessing how the patient's heart failure has prevented them from living the way they wanted during the defined time period. Each question was graded by the patient with a numeric value between 0 (No/none) and 5 (very much). These scores were then summed across the 21 questions for a Global Score. Global scores ranged from 0 to 105. These questions were further grouped into Physical (8 of the questions) and Emotional (5 of the questions) dimensions to further characterize the effect of heart failure on the patient's life. Physical scores ranged from 0 to 40, and emotional scores ranged from 0 to 25. For all 3 categories, the lower the score, the better the outcome. Values presented as change from Baseline.
Time Frame: 12 weeks
Population: Intention to treat population.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Inhaled Treprostinil | Placebo
Number analyzed (Participants) | 115 | 120
units on a scale
  Global Score | -3.0 (18.7) [-14.0 to 2.0] | 0.0 (16.2) [-9.0 to 6.0]
  Physical Dimension | -1.4 (8.9) [-6.0 to 2.0] | 0.0 (7.1) [-4.0 to 3.0]
  Emotional Dimension | 0.0 (5.7) [-4.0 to 1.0] | 0.0 (5.7) [-3.0 to 3.0]
Statistical Analysis 1: Comparison: Inhaled Treprostinil vs Placebo; Global Score; Test type: Superiority or Other; p = 0.027, Wilcoxon rank sum test; Hodges-Lehman Estimate = -4.0, 95% CI 2-sided [-8.0 to 0]
Statistical Analysis 2: Comparison: Inhaled Treprostinil vs Placebo; Physical Dimension; Test type: Superiority or Other; p = 0.037, Wilcoxon rank sum test; Hodges-Lehman Estimate = -2.0, 95% CI 2-sided [-3.0 to 0.0]
Statistical Analysis 3: Comparison: Inhaled Treprostinil vs Placebo; Emotional Dimension Score; Test type: Superiority or Other; p = 0.173, Wilcoxon rank sum test; Hodges-Lehman Estimate = -1.0, 95% CI 2-sided [-2.0 to 0.0]

8. Secondary Outcome: Change in Signs and Symptoms of PAH
Description: Signs and symptoms of PAH (Loud P2 sound, Ascites, Right ventricular S3 sound, Dyspnea, Right ventricular S4 sound, Orthopnea, Right ventricular heave, Dizziness, Murmur of tricuspid insufficiency, Syncope, Murmur of pulmonic insufficiency, Chest pain, Hepatomegaly, Palpitations, Jugular venous distension at 45 degrees, Fatigue, Edema) were assessed at Baseline and Week 12. The status of each sign and symptom ("absent" or "present") was assessed at each visit. To assess overall change from baseline in signs and symptoms, a "1" was assigned for each sign and symptom that was "present" at the Week 12 but was "absent" at baseline, a "-1" was assigned for each sign and symptom that was "absent" at Week 12 but was "present" at baseline, and a "0" was assigned for no change. An overall change score at each post-baseline assessment was then calculated by summing these values for all signs and symptoms. The overall change score had the potential to range from -17 to 17.
Time Frame: 12 weeks
Population: Intention to treat population.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Inhaled Treprostinil | Placebo
Number analyzed (Participants) | 115 | 120
units on a scale | 0 (3.5) [-6 to 5] | 0 (2.5) [-6 to 16]

9. Secondary Outcome: N-terminal Pro-B-Type Natriuretic Peptide (NT Pro-BNP)
Description: Change in NT pro-BNP from Baseline to Week 12. Plasma samples were collected from patients at Baseline and Week 12 in order to measure any change over time in circulating plasma levels of this biomarker.
Time Frame: 12 weeks
Population: Per protocol
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Inhaled Treprostinil | Placebo
Number analyzed (Participants) | 73 | 82
pg/mL
  Week 12 | 377 [124 to 1091] | 756 [177 to 2213]
  Change from Baseline | -57 [-396 to 34] | 40 [-93 to 288]
Statistical Analysis 1: Comparison: Inhaled Treprostinil vs Placebo; Test type: Superiority or Other; p = 0.001, Wilcoxon rank sum test; Hodges-Lehman Estimate = -167, 95% CI 2-sided [-333 to -64]

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Inhaled Treprostinil | Placebo
Serious Adverse Events (participants affected / at risk) | 9/115 | 13/120
Other Adverse Events (participants affected / at risk) | 101/115 | 100/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Treprostinil (N=115) | Placebo (N=120)
Worsening PAH (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Syncope (Nervous system disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diabetes mellitus (Endocrine disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
right ventricular failure (Cardiac disorders) | 1 | 0
Anxiety (Nervous system disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
blood potassium increased (Metabolism and nutrition disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Congestive cardiac failure (Cardiac disorders) | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
Cholelithiasis (Gastrointestinal disorders) | 0 | 1
Cor pulmonale (Cardiac disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Hematuria (Blood and lymphatic system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hypotension (Cardiac disorders) | 0 | 1
iron deficiency anemia (Metabolism and nutrition disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Treprostinil (N=115) | Placebo (N=120)
cough (Respiratory, thoracic and mediastinal disorders) | 62 | 35
headache (Nervous system disorders) | 47 | 27
dizziness (Nervous system disorders) | 20 | 18
nausea (Gastrointestinal disorders) | 22 | 13
throat irritation (Respiratory, thoracic and mediastinal disorders) | 16 | 10
Upper respiratory tract infection (Infections and infestations) | 10 | 14
fatigue (General disorders) | 10 | 12
diarrhea (Gastrointestinal disorders) | 11 | 9
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 7
flushing (Vascular disorders) | 17 | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 6
chest discomfort (General disorders) | 7 | 4
pain in jaw (Musculoskeletal and connective tissue disorders) | 6 | 5
nasopharyngitis (Infections and infestations) | 2 | 7
palpitations (Cardiac disorders) | 2 | 7
epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 2
syncope (Nervous system disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the United Therapeutics publication policy. The rights of the investigator and of the sponsor with regard to publication of the results are described in the investigator contract.